CLINICAL TRIAL: NCT01563185
Title: A Multicenter, Open-label Safety and Pharmacokinetic Study of DUEXIS® (Ibuprofen and Famotidine) Tablets in Juvenile Idiopathic Arthritis
Brief Title: Open-label Safety and Pharmacokinetic Study of DUEXIS® (Ibuprofen and Famotidine) Tablets in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Pediatric Rheumatology Collaborative Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ-CA-402
Record Dates: First submitted 2012-03-20; First posted 2012-03-26 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA; ibuprofen; famotidine; pediatrics; for > 1 month
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DUEXIS (Experimental): 800 mg ibuprofen/26.6 mg famotidine
  Interventions: Drug: 800 mg ibuprofen/26.6 mg famotidine

INTERVENTIONS:
Drug: 800 mg ibuprofen/26.6 mg famotidine — Oral tablet taken three time per day
  Other Names: DUEXIS

SUMMARY:
The primary objective of this Phase 4, multi-center, open-label study is to evaluate the safety and tolerability of DUEXIS in Juvenile Idiopathic Arthritis (JIA) patients aged 10 years to 16 years, 11 months, treated up to 24 weeks.

The secondary objectives are to evaluate the PK characteristics of DUEXIS in JIA patients and to evaluate the signs and symptoms of JIA in patients aged 10 years to 16 years, 11 months receiving DUEXIS for up to 24 weeks.

DETAILED DESCRIPTION:
Approximately 30 JIA patients who meet all eligibility criteria and who are expected to require daily administration of an NSAID for up to 24 weeks will be enrolled. A subset of approximately 6 patients will participate in a single dose PK study at Day 0 with an abbreviated PK profile performed at Week 4 if possible. Multiple dose PK sampling will occur in all enrolled patients.

Study with completed results acquired from Horizon in 2024

ELIGIBILITY:
Inclusion Criteria:

1. Patient and guardian are willing to consent to undergo up to 24 weeks of treatment with DUEXIS (ibuprofen 800 mg/famotidine 26.6 mg) oral tablet three times daily.
2. Patient is male or female, aged 10 years to 16 years, 11 months.
3. Patient is diagnosed with JIA for > 1 month including oligoarthritis, polyarthritis rheumatoid factor (RF) +, polyarthritis RF-, psoriatic arthritis, enthesitis-related arthritis, or undifferentiated and systemic arthritis without systemic features in the past 6 months.
4. Patient must have currently active articular disease as defined by > 1 active joint (i.e., presence of swelling, or if no swelling is present, limitation of motion [LOM] accompanied by pain, tenderness, or both).
5. Based upon investigator judgment, given current treatment patient is receiving and level of disease activity, it is determined appropriate for the patient to undergo up to 24 weeks of treatment with DUEXIS (ibuprofen 800 mg/famotidine 26.6 mg) oral tablet three times daily. The investigator will use his/her clinical judgment in determining the duration of treatment for the patient based on the standard of care up to 24 weeks of treatment.
6. Weight > 48 kg and body mass index (BMI) > 5th percentile using the Centers for Disease Control (CDC) BMI percentile calculator for child and teen at the screening visit.
7. Patient is able to swallow a DUEXIS tablet whole.
8. For the single dose pharmacokinetic (PK) subset, patients and guardians must be willing to participate in the serial blood sample collections at Day 0 and Week 4.
9. Female patients of childbearing potential and male patients must agree to use medically acceptable methods of contraception, including abstinence, throughout the entire study period.
10. Patient is willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

1. Patient has a history of or experienced any of the following:

   * NSAID-associated and/or primary peptic ulcer disease-associated serious gastrointestinal complications such as perforation of ulcers, gastric outlet obstruction due to ulcers, and/or acute gastrointestinal bleeding
   * NSAID-induced asthma exacerbation, acute renal failure, interstitial nephritis, and/or hepatitis
   * Malignant disease of the gastrointestinal tract
   * Erosive esophagitis
   * Coronary artery bypass graft (CABG) surgery within the 14 days prior to study Day 0
   * Uncontrolled diabetes mellitus as evidenced by Hemoglobin A1c > 7%
   * Known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C.
2. Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral disease.
3. JIA disease is severe as defined by either physician's or parent's global assessments > 90 on a 100 point scale.
4. Systemic JIA with any of the following manifestations within the last 6 months prior to enrollment: intermittent fever due to JIA, rheumatoid rash, hepatosplenomegaly, pleuritis, pericarditis, or macrophage activation syndrome.
5. Active uveitis.
6. Presence of any other rheumatic disease or major chronic infectious, inflammatory, immunologic disease (e.g., inflammatory bowel disease, hypogammaglobulinemia, or systemic lupus erythematosus, etc.).
7. Presence at screening or history of any disease other than JIA that requires the use of chronic systemic corticosteroids.
8. History of clinically significant drug or alcohol abuse.
9. Presence at screening of any of the following laboratory values:

   * Hemoglobin < 9.0 g/dL
   * White blood cells < 2000/mm^3 (2 x 109/L)
   * Platelets < 150,000/mm^3 (150 x 109/L)
   * Serum creatinine > 1.5 times upper limit of normal
   * Serum ALT or AST > 2.0 times upper limit of normal
   * H. pylori positive
   * Any other lab value that in the opinion of the investigator might place the patient at unacceptable risk for participation in this study.
10. Methotrexate > 20 mg/M^2/week or > 40 mg/week.
11. Patient currently is participating in an investigational drug study, or patient participated in an investigational drug study within the 30 days (or < 5 terminal half-lives of elimination) prior to study entry.
12. Females who are pregnant or breast feeding.
13. Female patient has a positive serum pregnancy test at Screening and/or a positive urine pregnancy test at Study Day 0.
14. Patient has a concomitant disease or condition that, in the opinion of the Investigator, could interfere with the conduct of the study or could put the patient at unacceptable risk

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Children's Hospital, New Orleans, Louisiana
  - Floating Hospital for Children @ Tufts Medical Center, Boston, Massachusetts
  - UMASS Memorial Children's Medical Center, Worcester, Massachusetts
  - Altoona Center for Clinical Research Altoona Arthritis, Duncansville, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DUEXIS
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-Compliance with study drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs)
Description: Safety assessments included AE monitoring, concomitant medication review, physical examinations (including vital signs and weight), and clinical laboratory assessments, including pregnancy testing for female patients. The outcome measure data table below describes the TEAEs experienced by patients.
Time Frame: Day 0 through Week 26/ET (adverse event data was collected at every visit, including telephone visits)
Measure: Number; unit: participants
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
participants
  Any patient with at least 1 TEAE | 12
  Any patient with at least 1 mild TEAE | 7
  At least 1 moderate TEAE | 5
  At least 1 severe TEAE | 0
  A possibly related TEAE | 2
  SAE | 0
  A TEAE leading to study drug discontinuation | 0
  A TEAE leading to death | 0
  TEAE: Gastrointestinal Disorders | 4
  TEAE: General disorders | 2
  TEAE: Infections and infestations | 7
  TEAE: Injury, poisoning & procedural complications | 2
  TEAE: Muscoskeletal & connective tissue disorders | 2
  TEAE: Nervous system disorders | 1
  TEAE:Respiratory, thoracic & mediastinal disorders | 3
  TEAE: Skin and subcutaneous tissue disorders | 2

2. Secondary Outcome: Childhood Health Questionnaire Parent Form 50 (CHQ-PF50) Scores
Description: To assess patient quality of life while on study medication, the CHQ was administered to the patients' parent or guardian on Day 0 and at the Week 24/ET visit. The raw scale scores were transformed into scores on a 0 to 100 scale, 100 indicating best health and 0 indicating worst health. The algorithm is:
  Transformed Score = ((Actual Raw Score - Lowest Possible Raw Score)/(Possible Raw Score Range)) x100. The actual raw score is the mean of the item responses in a scale (sum of item responses/number of completed items). The possible raw score range is the highest possible raw score minus the lowest possible raw score. The outcome measure data table shows the average change in the CHQ concepts from Baseline to the week 24 visit. The average change in the CHQ concepts is on a -100 to 100 scale, -100 representing a negative change in health and 100 indicating a positive change in health.
Time Frame: Baseline to Endpoint (Endpoint is the last post-baseline value obtained, as two subjects did not complete the study up until week 24).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
units on a scale
  Global Health | 2.5 (21.16)
  Physical Functioning | 19.0 (36.29)
  Role/Social Limitations: Emotional/Behavioral | 14.8 (35.86)
  Role/Social Limitations: Physical | 20.8 (32.68)
  Bodily Pain/Discomfort | 15.8 (27.12)
  Behavior | 8.4 (13.29)
  Global Behavior Item | 6.7 (10.30)
  Mental Health | 3.3 (9.37)
  Self Esteem | 5.3 (12.47)
  General Health Perceptions | 1.9 (14.40)
  Change in Health | 14.6 (39.11)
  Parental Impact: Emotional | 20.4 (24.51)
  Parental Impact:Time | 22.2 (30.92)
  Family Activities | 14.3 (26.80)
  Family Cohesion | 4.6 (8.65)

3. Secondary Outcome: American College of Rheumatology (ACR) Pediatric Core Measures: Physician's Global Assessment of Disease Activity and Parent's Assessment of Overall Well-being
Description: The following 2 ACR pediatric Core Measures of JIA activity and the parent's assessment of discomfort were quantitatively assessed at baseline and each study visit: the physician's global assessment of disease activity and the parent's global assessment of overall well-being. These ACR values represent the average change in the physician's global assessment of disease activity and the parent's global assessment of overall well-being from the baseline visit to the week 24/ET visit. The ACR pediatric core measure: Physician's global assessment of disease activity and parent's assessment of overall well being was measured on a scale of 0-100 mm (0 = very good, 100=very poor).
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
units on a scale
  Physician's Global Assessment of Disease Activity | -9.1 (28.34)
  Parent's Global Assessment of Overall Well-Being | -8.0 (34.07)

4. Secondary Outcome: American College of Rheumatology (ACR) Pediatric Core Measures: CHAQ - Disability Index
Description: The following ACR pediatric Core Measure of JIA activity and the parent's assessment of discomfort were quantitatively assessed at baseline and each study visit: CHAQ - Disability Index. This ACR measurement represents the average change in the Childhood Health Assessment Questionnaire (CHAQ) - Disability Index from the baseline visit to the week 24/ET visit. The CHAQ disability index is measured on a scale of 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do).
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
units on a scale | -0.146 (0.3235)

5. Secondary Outcome: ACR Pediatric Components by Time Point: Number of Joints With Active Arthritis and the Number of Joints With Limited Range of Motion Number of Joints With Active Arthritis
Description: The following 2 ACR pediatric Core Measures of JIA activity and the parent's assessment of discomfort were quantitatively assessed at baseline and each study visit: number of joints with active arthritis and the number of joints with limited range of motion. These ACR values represent the average change in number of joints with active arthritis and the number of joints with limited range of motion from the baseline visit to the week 24/ET visit.
  The joints that were assessed include the right and left temporomandibular, sternoclavicular, arcomiclavicular, shoulder, elbow, wrist, MCP - 1. MCP - 2, MCP - 3, MCP - 4, MCP - 5, PIP - 1, PIP - 2, PIP - 3, PIP - 4, PIP - 5, DIP - 1, DIP - 2, DIP - 3, DIP - 4, and DIP - 5.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: Number of joints
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
Number of joints
  Number of joints with active arthritis | -4.3 (6.97)
  Number of joints with limited range of motion | -1.7 (5.43)

6. Secondary Outcome: American College of Rheumatology (ACR) Pediatric Core Measures: Serum C Reactive Protein (CRP) Concentration
Description: The following ACR pediatric Core Measure of JIA activity and the parent's assessment of discomfort were quantitatively assessed at baseline and each study visit: CRP Concentration. This ACR value represents the average change in Serum C Reactive Protein (CRP) Concentration from the baseline visit to the week 24/ET visit. The normal range referenced was 0 mg/L - 4.99 mg/L.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | DUEXIS
Number analyzed (Participants) | 12
mg/L | 1.019 (3.9742)

7. Secondary Outcome: Single Dose Pharmacokinetic Characteristics of DUEXIS in JIA Patients: Time of Maximum Observed Concentration (Tmax)
Description: Tmax was estimated for ibuprofen and famotidine.The PK parameters for ibuprofen and famotidine represent average Tmax values following a single oral dose of DUEXIS. Samples were collected pre-dose and at 0.5, 1, 2, 4, and 8 to 10 hours following study drug administration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8 hours post-dose
Population: The initial 9 patients met the PK objective of the study (4 were in the single dose pharmacokinietic group, however, 1 of the patients was not evaluable, and all 9 were in the multiple dose pharmacokinetic group).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DUEXIS
Number analyzed (Participants) | 3
hours
  Tmax: Ibuprofen | 1.75 (0.66)
  Tmax: Famotidine | 2.1 (0.14)

8. Secondary Outcome: Single Dose Pharmacokinetic Characteristics of DUEXIS in JIA Patients: Maximum Observed Concentration (Cmax)
Description: Cmax was estimated for ibuprofen and famotidine. The PK parameters for ibuprofen and famotidine represent average Cmax values following a single oral dose of DUEXIS. Samples were collected pre-dose and at 0.5, 1, 2, 4, and 8 to 10 hours following study drug administration.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DUEXIS
Number analyzed (Participants) | 3
ug/mL
  Cmax: Ibuprofen | 49.8 (13.7)
  Cmax: Famotidine | 55.0 (11.9)

9. Secondary Outcome: Single Dose Pharmacokinetic Characteristics of DUEXIS in JIA Patients: Area Under the Concentration-time Curve From the Time of Dosing to the Last Measurable Concentration (AUC(0-t))
Description: AUC(0-t) was estimated for ibuprofen and famotidine. The PK parameters for ibuprofen and famotidine represent average AUC values following a single oral dose of DUEXIS. Samples were collected pre-dose and at 0.5, 1, 2, 4, and 8 to 10 hours following study drug administration.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8 hours post-dose
Population: The initial 9 patients met the PK objective of the study (4 were in the single dose pharmacokinietic group, however, 1 patient was not evaluable, and all 9 were in the multiple dose pharmacokinetic group).
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | DUEXIS
Number analyzed (Participants) | 3
ug*h/mL
  AUC(0-t): Ibuprofen | 196.5 (27.4)
  AUC(0-t): Famotidine | 267.6 (27.1)

10. Secondary Outcome: Multiple Dose Pharmacokinetic Characteristics of DUEXIS in JIA Patients: Individual Oral Clearance (CL/F)
Description: CL/F was estimated in ibuprofen and famotidine.
Time Frame: Pre-dose and 0.5, 1, 2, 4, and 8 hours post-dose in the single dose group; sparse samples at random times in the multiple dose group
Population: The initial 9 patients met the PK objective of the study (4 were in the single dose pharmacokinietic group, however, 1 of the patients was not evaluable and all 9 were in the multiple dose pharmacokinetic group).
Measure: Mean (Standard Deviation); unit: L/h/70 kg
Arm/Group | DUEXIS
Number analyzed (Participants) | 9
L/h/70 kg
  CL/F: Ibuprofen | 2.8 (0.6)
  CL/F: Famotidine | 61.5 (15.9)

11. Secondary Outcome: Multiple Dose Pharmacokinetic Characteristics of DUEXIS in JIA Patients: Volume Distribution (V/F)
Description: V/F were estimated in ibuprofen and famotidine.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/70 kg
Arm/Group | DUEXIS
Number analyzed (Participants) | 9
L/70 kg
  V/F: Ibuprofen | 16.7 (4.6)
  V/F: Famotidine | 564.4 (154.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the Day 0 visit up until the Follow-up visit (Week 26). Adverse events were collected at the following time points: Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 26.
Arm/Group | DUEXIS
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DUEXIS (N=12)
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral viral infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less